CLINICAL TRIAL: NCT01240473
Title: A Pilot Study for Capacity Building for a Multi-centre, Randomized Trial for Treatment of Kala Azar in Bangladesh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Community Based Medical College, Bangladesh (Other); Dhaka Medical College (Other); Directorate General of Health Services of Bangladesh (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-008; 2007-008
Record Dates: First submitted 2010-11-07; First posted 2010-11-15 (Estimated); Last update posted 2018-03-16 (Actual); Status verified 2010-11

CONDITIONS: Visceral Leishmaniasis
Keywords: kala azar; visceral leishmaniasis; diagnosis; drug resistance; Therapeutics; Capacity Building
MeSH Terms: conditions — Leishmaniasis, Visceral; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Randomized trial for treatment of kala azar in Bangladesh — dose of SAG 20 mg/kg body weight, with a maximum dose of 850 mg/day, for 28 days

SUMMARY:
Kala azar (KA) or visceral leishmaniasis (VL) is endemic in several districts of Bangladesh with the highest incidence in Mymensingh, Pabna and Tangail districts. ICDDR,B is involved in a project for improving the surveillance of KA in Trishal, Mymensingh since 2005. Improvement of case detection is necessary for both surveillance purposes and better control. The aims of this pilot study are to assess some newer techniques for diagnosis of KA using blood and urine samples of suspected cases; and evaluate response to treatment with sodium stibogluconate to which resistance has been reported in India, considered to be a part of the same zone harboring the disease agent Leishmania donovani and transmitted by the same vector Phlebotomas argentipes (sand-fly). No data is currently available on response to sodium stibogluconate in KA patients in Bangladesh. Although a number of new drugs have been evaluated in the treatment of KA in India and Kenya, no trial has so far been conducted in Bangladesh. A team of researchers from GlaxoSmithKline (UK) had recently visited Bangladesh to evaluate if it would be possible to conduct a Phase-III clinical trial with sitamaquine. They interacted with scientists of ICDDR,B and expressed their interest to help develop ICDDR,B's capacity in order to include Bangladesh as one of the sites for the planned, multi-centre, Phase-III trial of sitamaquine; India and Nepal are two other possible sites for the trial. The aims of the proposed study are to train physicians and laboratory personnel in preparation for the future drug trial(s) on KA as well as to compare different tests for its diagnosis that might improve case detection at the field level and used for research purposes. The investigators will also examine in greater detail the different Leishmania species circulating in the area of Mymensingh and whether treatment failure and occurrence of Post Kala azar Dermal Leishmaniasis (PKDL) is associated with certain species.

DETAILED DESCRIPTION:
Specific Aims:

Primary objective: To develop capacity to evaluate newer regimens for treatment of kala azar in Bangladesh.

Secondary objectives:

1. To evaluate novel diagnostic tests for kala azar including rK39 dipstick test in serum; KATEX in urine; and PCR (polymerase chain reaction) in blood and clinical samples.
2. To evaluate response to treatment with 28 injections of SAG using PCR in blood samples and clinical samples.
3. To transfer the mini-exon PCR-RFLP technique to ICDDR,B and to characterize the most prevalent Leishmania species in the area of Mymensingh and their response to standard treatment with SAG.
4. We will also analyze whether certain genotypes are associated with the occurrence of PKDL and whether the mini-exon PCR is a suitable marker for monitoring the intra and interspecies genetic evolution of Leishmania species.

Research Design and Methods:

The patients for the proposed study were selected from three upazilla health complexes in Mymensingh per discussion with the government agencies working in these areas. If necessary, we would go for active surveillance to enroll required number of subjects for the study.

Patients

In total, 200 consecutive cases (age >5 years) meeting the following diagnostic criteria for KA were enrolled into the study: (i) fever for >2 weeks; (ii) at least one of the the following criteria- splenomegaly, darkening of the skin, and weight loss; and (iii) a positive rK39 dipstick test. Exclusion criteria will include: (1) children under five years of age, (2) pregnant women, and (3) patients who are suffering simultaneously from any other serious illness which is unrelated to kala azar. Patients (or their parents/guardians in the event of minors) meeting the above criteria, was explained about the risk of treatment with SAG and the risk involved in splenic aspiration procedures by expert physicians. Informed consent (verbal or written) was then obtained from the patients (or their parents/guardians in the event of minors) before inclusion into the study. One hundred healthy individuals living in the same area were enrolled as controls for evaluating PCR and other diagnostic tests of KA. Our field workers visited houses in the community and collect blood samples from the healthy volunteers with their informed consent.

Study procedures and assessments

Splenic aspiration:

Splenic aspiration was performed in 200 consecutive patients who had been presented with clinical features of KA with a positive rK39 dipstick test. Splenic aspiration was performed for confirmation of diagnosis on study day 1, and then again on day 29 to assess cure from the disease. Thus, when a subject was found to be positive by rK39 dipstick test, standard pre-procedure tests for splenic aspiration e,g. hemoglobin estimation, bleeding time, clotting time, and platelet counts, were performed. Splenic aspiration was performed only in those who were not severely anemic (Hb ≥ 6 mg/dl), and had platelet counts of >50,000/micro liter of blood. Prothrombin time was also be checked before splenic aspiration and those with a PT more than 4 seconds prolonged were not be eligible for the study. All necessary treatment was provided in the event of hemorrhage following the procedure, including blood transfusion. If necessary, the patients also be transported to Mymensingh Medical College Hospital, for more specialized treatment and support.

Treatment and follow up

In Bangladesh, intramuscular administration of sodium antimony gluconate (SAG; Albert David Ltd., India), in a dose of 20 mg/kg body weight, with a maximum dose of 850 mg/day, for twenty eight days is the current standard treatment for patients with KA. The pulse and respiratory rates, blood pressures, and temperature were monitored at 12 hourly intervals during this treatment period. EKG were performed if clinically indicated. The treatment was stopped if signs of severe toxicity (cardiotoxicity, renal failure, etc) develop, and the patient had been treated with standard dose of amphotericin B.

Hospitalization: All patients under treatment was offered to stay at Community-based Medical College Hospital for the entire period of treatment with SAG. The patients had been hospitalized for treatment with amphotericin B in case of treatment failure or toxicity with SAG.

Follow up: At the end of treatment, the patients was evaluated for cure by physical examination and splenic aspiration. The subjects had been following for six months as shown in Scheme-2.

Diagnostic tests to be evaluated

rK39 dipstick test A finger-prick blood specimen was collected in capillary tubes for rK39 dipstick test. This method is rapid and time saving.

Parasitological diagnosis

Splenic aspirate was used for parasitological diagnosis. A slide of splenic aspirates was prepared for Giemsa staining. Two lab technicians from ICDDR,B was trained on staining techniques and reading of the slides. Randomly selected slides had been sent to reference labs elsewhere for Quality Control.

Polymerase chain reaction (PCR)

DNA of Leishmania donovani in the collected blood samples had been detected using the methods described by Salotra et al.

Sample collection and DNA isolation: Collected blood specimen was transported to the Parasitology Laboratory of ICDDR,B, and transferred to 4°C and processed generally on the same day. DNA was extracted from 0.2 ml of blood using a QIAamp DNA blood mini kit (Qiagen).

PCR amplification: DNA from cultured parasites (1 ng) and from clinical samples (100 ng) were taken for amplification using the LdI primers described above. The reaction mixture (50 µl) contained 10 mM Tris-HCl (pH 8.3) 50 mM KCl, 1.5 mM MgCl2, a 200 µM concentration of each deoxynucleoside triphosphate, 50 ng of each primer, and 1.25 U of Taq DNA polymerase (Gibco BRL). Each reaction mixture was overlaid with mineral oil, and amplification was performed in a thermal cycler (Perkin-Elmer, Warrington, Great Britain) programmed for 40 cycles of denaturation at 94°C for 1 min, annealing at 45°C for 1 min, and extension at 72°C for 2 min, preceded by an initial denaturation of 2 min at 94°C. Final extension was for 3 min at 72°C. Products was analyzed by electrophoresis in 1% agarose gel containing ethidium bromide (0.5 µg/ml) in TAE buffer (0.04 M Tris acetate, 0.001 M EDTA) and photographed under UV illumination.

Mini-exon PCR-RFLP: The mini-exon PCR-RFLP had been developed by the Swiss Tropical Institute (STI) (Marfurth et al. 2003).

Sample Size Calculation and Outcome Variable(s):

The sample size of 200 cases and 100 controls is based on practical considerations for meeting the primary objective of capacity development and the study is not formally powered for hypothesis testing. The emphasis for investigating sensitivity and specificity of the new diagnostic tests will be on presenting descriptive statistics and confidence intervals.

Data Analysis:

The sensitivity (proportion of correctly identified true positive results) and specificity (proportion of correctly identified true negative results) was calculated for each diagnostic test, and 95% confidence intervals for these proportions had been calculated using Wilsons method.

The positive and negative predictive values was also be calculated using the method described by Altman et al. The positive predictive value is the proportion of patients with a positive result for the experimental diagnostic test who are correctly diagnosed by parasitological examination. Similarly the negative predictive value is the proportion of patients with a negative diagnostic test result who are correctly diagnosed by parasitological examination. The 95% CI for the positive and the negative predictive values had been determined. These parameters would allow the comparison of each diagnostic test with the 'gold standard' parasitological examination.

ELIGIBILITY:
Inclusion Criteria:

* KA will be enrolled into the study:

  * fever for >2 weeks
  * at least one of the the following criteria- splenomegaly, darkening of the skin, and weight loss
  * a positive rK39 dipstick test.

Exclusion Criteria:

* children under five years of age\
* pregnant women
* patients who are suffering simultaneously from any other serious illness which is unrelated to kala azar (for example, tuberculosis, cancer, etc).

Ages: 5 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2007-04; Primary Completion 2008-03 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
To develop capacity to evaluate newer regimens for treatment of kala azar in Bangladesh. | 1 year

SECONDARY OUTCOMES:
To evaluate response to treatment with 28 injections of SAG | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kazi M Jamil, MD, PhD, Principal Investigator — Associate Scientist
Locations (1):
- Community-based Medical College, Bangladesh (CBMC,B), Mymensingh, Dhaka Division, Bangladesh